CLINICAL TRIAL: NCT00463996
Title: Værdien af MRI Til Staging af c.Ovarii-et Prospektivt Studie
Brief Title: MRI in Staging Ovarian Cancer Using MRI Contrast Agent
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Aarhus (Other)
Other Study IDs: MR-Center-001
Record Dates: First submitted 2007-04-18; First posted 2007-04-20 (Estimated); Last update posted 2007-04-20 (Estimated); Status verified 2007-04

CONDITIONS: Ovarian Cancer
Keywords: Ovarian cancer; MRI; Contrast agent
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Can MRI be used to stage ovarian cancer?

DETAILED DESCRIPTION:
Staging of ovarian cancer can best be performed with CT or MRI compared to ultrasound. Studies have shown an increase in pos. predictive value by adding contrast i.v. to the MR-examination protocol. We compare staging of ovarian cancer by 1.MRI without contrast (standard method) to 2.MRI with contrast agent i.v. (new method)in the same patient. Golden standard are findings at operation.

ELIGIBILITY:
Inclusion Criteria:

* suspicion of ovarian cancer

Exclusion Criteria:

* recurrence of disease
* contraindication to MRI, contrast agent
* inoperable patients for other reasons

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50
Dates: Start 2007-04; Study Completion 2008-04 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Liselotte Ibsen, doc, Principal Investigator — Aarhus University Hospital, BDA, Skejby